CLINICAL TRIAL: NCT04262414
Title: Restoring Upright Mobility After Spinal Cord Injury Using Functional Electrical Stimulation
Brief Title: Restoring Upright Mobility After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-5151
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2020-02

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases
Keywords: Balance; Functional Electrical Stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Functional Electrical Stimulation — The device used was a prototype closed-loop FES system to improve standing balance by activating the ankle plantar flexors and dorsiflexors (i.e. A-FES system). As a closed-loop system, the body's position and velocity are continually monitored, and the level of stimulation adjusted accordingly on a moment-to-moment basis. This differs from currently available FES units, which do not monitor body movement and therefore, provide a constant level of stimulation unless manually adjusted by the user/PT. The control strategy used in the A-FES system mimics the physiological control system in able-bodied people, meaning it has the potential to "re-educate" normal movement patterns.

SUMMARY:
Up to 15 able-bodied individuals will participate in one testing session to evaluate the effectiveness of the A-FES system. Up to 20 individuals with SCI will participate in 12 sessions of A-FES therapy. At each session, participants will stand on a force plate (Accu Sway, AMTI, USA) with the A-FES system (Compex Motion II, Compex Motion, Switzerland) donned. The centre of pressure (COP) will be calculated in real time using the force plate data. The calculated COP will be presented to participants on a monitor and they will be instructed to shift their COP in the indicated directions as represented by a cursor (i.e. training with visual feedback). The intensity of electrical stimulation provided by the A-FES system will be regulated by the measured COP in a closed-loop manner. In this study we propose to develop and evaluate the clinically-feasible A-FES system for the training of standing balance.

ELIGIBILITY:
Inclusion Criteria:

1. A traumatic or non-traumatic, non-progressive (AIS) C or D SCI;
2. ≥18 years old;
3. Able to stand independently for 60s;
4. Moderate level of trunk control as evidenced by the ability to reach forward >2 inches in standing (i.e. score of 2 on the BBS Reaching Forward task50,51); and
5. Free of any other condition besides SCI that significantly affects walking or balance (e.g., no vestibular disorder, significant vision loss, stroke).

Exclusion Criteria:

1. Severe spasticity in the legs;
2. Contractures in the lower extremities that prevent achieving a neutral hip and ankle position, or extended knee;
3. A prior lower extremity fragility fracture;
4. An injection of botulinum toxin to leg muscles in the past six months;
5. Peripheral nerve damage in the legs (i.e. leg muscles unresponsive to electrical stimulation);
6. A pressure sore (>grade 2) on the pelvis or trunk where the safety harness is applied; o
7. Contraindications for FES52 (i.e. implanted electronic device, active cancer or radiation in past 6 months, epilepsy, skin rash/wound at a potential electrode site).

Participants will be withdrawn from the study if FES irritates their skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Change from Baseline Berg Balance Scale at 8 weeks
  Assesses static and dynamic standing balance; score 0-56; higher score means a better outcome
Mini-Balance Evaluation Systems Test | Change from Baseline Mini-Balance Evaluation Systems Test at 8 weeks
  Assesses four balance control systems, including anticipatory balance, reactive postural control, sensory orientation and dynamic gait
Activities-specific Balance Confidence Scale | Change from Baseline Activities-specific Balance Confidence Scale at 8 weeks
  A measure of balance self-efficacy; mean score of 0-100; higher score means a better outcome (i.e. high balance confidence)

SECONDARY OUTCOMES:
Static standing balance | Through study completion, average of 8 weeks
  Postural sway during quiet standing
Dynamic standing balance | Through study completion, average of 8 weeks
  Assessed by asking participants to lean as far as possible in the forward, backward and sideways directions while standing on a force plate (i.e. limits of stability test)
Semi-structured interview | up to 8 weeks post-intervention
  The guide will include open-ended questions concerning the participant's experience with, and impressions of, A-FES therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kristin E Musselman, PhD, Principal Investigator — University of Toronto
Locations (1):
- Lyndhurst Centre, Toronto Rehabilitation Institute-UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Houston DJ, Unger J, Lee JW, Masani K, Musselman KE. Perspectives of individuals with chronic spinal cord injury following novel balance training involving functional electrical stimulation with visual feedback: a qualitative exploratory study. J Neuroeng Rehabil. 2021 Apr 1;18(1):57. doi: 10.1186/s12984-021-00861-z. PMID 33794948